CLINICAL TRIAL: NCT00822562
Title: Research on Surgery and Micro-Invasive Treatment in Recurrent Primary Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-016; ZD2008-016-P1
Record Dates: First submitted 2009-01-06; First posted 2009-01-14 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procedure/Surgery (Active Comparator): surgery
  Interventions: Procedure: surgery
- Procedure (Experimental): PRFA or PMCT
  Interventions: Other: PRFA or PMCT

INTERVENTIONS:
Other: PRFA or PMCT — PRFA or PMCT 30-35W for 10-15minutes one cycle,three cycles
  Arms: Procedure
Procedure: surgery — only surgery
  Arms: Procedure/Surgery

SUMMARY:
In this study, we intend to divide the subjects who have been confirmed recurrent HCC into two groups: Group A: treatment with pure surgery or Group B: treatment with pure radio frequency. We will compare the non-tumor survival time, long-term survival rate between the two groups, summarize the merits and demerits of both groups, and try to establish a standardized therapy and treatment for the this kind of patients through prospective studies on the molecular biological difference of pathological samples between the first and second surgeries.

DETAILED DESCRIPTION:
The recurrence and metastasis of primary liver cancer (PLC) have always been a tough problem for surgeons. Gu Hong-guang reported the five years recurrence rate in PLC subjects reached 75~100%, among which 60% were discovered within three years after surgeries, with the peak appearing at 18~24 months. According to a report delivered by Zhong-Shan Hospital, the recurrence rate of small HCC was 40%, and that of large HCC was 1.9 times of small HCC. Chen Han agreed that the recurrence rate in 1~2 years reached 71.6%, while in 2~11 years was 28.4%. With the rapid development of iconography and surgical techniques, it is possible for surgeon to resect the recurrent HCC now. In 1986, Nagasue et al. reported the excision of recurrent HCC and proved that comparing with non-surgical treatment, subjects with recurrent HCC excision got a higher survival rate. However, the excision rate of recurrent HCC has always been an arguable point. Nakajima et al. suggested the excision rate in 133 subjects was 24%, while Matsuda et al. agreed that in 91 subjects reached 44%, and Zhoo reported that in 384 subjects was 35%; Kakazu et al. insisted that in 286 subjects was 17%; Nagasue et al. said that in 290 subjects was 30%; Shoto et al. reported that in 341 subjects was 19% and Poon et al. advocated that in 244 subjects was 10%. He Sheng summarized the 1295 subjects in recent five years, and only 106 of them had the opportunities to have excision again (8.18%). Sugimachi, Minagawa et al. reported separately the 5 year survival rate in recurrent HCC subjects were 47.5% and 56.0%, which showed no significant difference with the first surgeries, but better therapeutic effects, meanwhile, third and forth surgeries could also get similar survival rate, which indicated that surgical excision is a vital treatment in recurrent HCCs. Chen Han in our hospital reported the first, third, fifth, and tenth year survival rate in 162 recurrent HCC subjects who underwent first surgical treatment were separately 96.8%, 66.7%, 43.6% and 21.8%; while that in subjects who received second surgical treatment were separately 94.7%, 44.9% and 25.0% at the first, third, and fifth year (mean survival time was 45 months, and average survival time was 54 months).

In this study, we intend to divide the subjects who have been confirmed recurrent HCC into two groups: Group A: treatment with pure surgery or Group B: treatment with pure radio frequency. We will compare the non-tumor survival time, long-term survival rate between the two groups, summarize the merits and demerits of both groups, and try to establish a standardized therapy and treatment for the this kind of patients through prospective studies on the molecular biological difference of pathological samples between the first and second surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. 20~60 years old;
2. diagnosed HCC pathologically, and confirmed recurrent HCC through ultrasonic B, CT, MRI or DSA test;
3. has a good condition in vital organs such as heart, lung, and kidney;
4. has a good liver function: Child A level, or nearly A level after hepatoprotection treatment;
5. solitary small cancer focus (diameter <5cm), or the number of recurrent HCC focus is no more than three and all of them grow in the same lobe of liver;
6. without jaundice (not including jaundice in the bile ducts), without ascites or extensive metastasis outside the liver;
7. without invasion to portal vein.

Exclusion Criteria:

1. subjects refuse to participate in this study;
2. subjects cannot be followed up regularly;
3. subjects with severe heart, lung, kidney diseases;
4. subjects with liver CP level B or C, and serum creatinine ≥2×ULN;
5. subjects with severe bone marrow depression, such as neutrophil counting is lower than 1.5 × 109.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | two years

SECONDARY OUTCOMES:
non-tumor life span, intra-liver recurrence rate, metastasis rate | two years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital Affiliated to Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xia Y, Li J, Liu G, Wang K, Qian G, Lu Z, Yang T, Yan Z, Lei Z, Si A, Wan X, Zhang H, Gao C, Cheng Z, Pawlik TM, Wang H, Lau WY, Wu M, Shen F. Long-term Effects of Repeat Hepatectomy vs Percutaneous Radiofrequency Ablation Among Patients With Recurrent Hepatocellular Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2020 Feb 1;6(2):255-263. doi: 10.1001/jamaoncol.2019.4477. PMID 31774468